CLINICAL TRIAL: NCT06016881
Title: Prospective Observational Study of Postoperative Chronic Operation-related Symptoms and Long-term Survival Quality After Minimally Invasive Lung Surgery
Brief Title: Postoperative Chronic Operation-related Symptoms After Minimally Invasive Lung Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POSLS-union01
Record Dates: First submitted 2023-08-21; First posted 2023-08-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer Stage I; Quality of Life
Keywords: lung cancer; Surgery; Quality of Life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer has been the most commonly diagnosed cancer globally over the past few decades. Histologically, adenocarcinoma in situ (AIS) and minimally invasive adenocarcinoma (MIA) are defined as cancers with no or limited tissue infiltration. Studies have shown that patients with AIS or MIA have a 100% probability of being free of recurrence within 5 years after surgery and have disease-specific survival rates of 100% and 100%, respectively.

In patients with early-stage lung cancer and benign lesions, long-term postoperative survival and tumor recurrence are non-priorities. Therefore, perioperative and postoperative quality of life are increasingly emphasized by patients and clinicians. However, a significant proportion of patients undergoing minimally invasive lung surgery still develop chronic pain and chronic cough in the postoperative period, the severity of which can lead to reduced quality of life. In addition, studies of the psychological state of patients undergoing surgery for pulmonary nodules are rare, and we believe this is one of the valuable factors affecting quality of life. The investigators have launched the first prospective observational trial to investigate the incidence of long-term chronic symptoms after minimally invasive lung surgery, risk factors, treatment received and treatment efficacy, duration of disease, and eventual regression, in addition to pre- and postoperative psychological status and long-term postoperative quality of life in patients undergoing minimally invasive lung surgery.

DETAILED DESCRIPTION:
Lung cancer has been the most commonly diagnosed cancer globally over the past few decades. With the widespread use of Low-dose computedtomograph (LDCT), more and more lung nodules are being detected. With the exception of benign nodules, the vast majority of lung cancer nodules are early stage lung cancers with predominantly ground glass lesions. Histologically, adenocarcinoma in situ (AIS) and minimally invasive adenocarcinoma (MIA) are defined as cancers with no or limited tissue infiltration. Studies have shown that patients with AIS or MIA have a 100% probability of being free of recurrence within 5 years after surgery and have disease-specific survival rates of 100% and 100%, respectively.

In patients with early-stage lung cancer and benign lesions, long-term postoperative survival and tumor recurrence are non-priorities. Therefore, perioperative and postoperative quality of life are increasingly emphasized by patients and clinicians. Enhanced rapid recovery management after video-assisted thoracoscopic surgery (VATS) can minimize the damage and impact of surgery on patients. However, a significant proportion of patients undergoing minimally invasive lung surgery still develop chronic pain and chronic cough in the postoperative period, the severity of which can lead to reduced quality of life. In addition, studies of the psychological state of patients undergoing surgery for pulmonary nodules are rare, and we believe this is one of the valuable factors affecting quality of life. The investigators have launched the first prospective observational trial to investigate the incidence of long-term chronic symptoms after minimally invasive lung surgery, risk factors, treatment received and treatment efficacy, duration of disease, and eventual regression, in addition to pre- and postoperative psychological status and long-term postoperative quality of life in patients undergoing minimally invasive lung surgery.

The researchers included patients with stage I lung cancer and benign lesions who underwent single-port thoracoscopic lung surgery. Patients' baseline levels, including usual chronic pain, chronic cough, and sleep, were recorded prior to surgery, and anxiety, depression, and quality of life scores were performed using the Generalized Anxiety Disorder Screener (GAD-7), Beck Depression Inventory (BDI), Hospital Anxiety and Depression Scale (HADS), and the European Organisation for Research and Treatment of Cancer (EORTC) 30 item Quality of Life Questionnaire (QLQ-C30). For the first 3 days after surgery, Pain, cough, nausea and vomiting were assessed using the numeric pain rating scale (NRS) and the visual simulation scale (VAS) score 3 times a day (every 8 hours), and sleep status were recorded each day. Anxiety and depression were evaluated during postoperative hospital stay. Postoperative chronic symptoms and quality of life will be assessed at postoperative weeks 1, 2, 4, 12, 26, and 52. Chronic cough will be assessed using the Leicester Cough Questionnaire, chronic pain will be assessed using Brief Pain Inventory and McGill Pain Questionnaire, and EORTC QLQ-C30 questionnaire, HADS, GAD-7 and BDI for continuous assessment of quality of life, anxiety status and depression status, as well as to record the time of onset of chronic symptoms, predisposing factors, aggravating and relieving factors, the presence or absence of treatment, the effectiveness of the treatment, and time of exacerbation, remission or disappearance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above;
2. Received single-port thoracoscopic surgery;
3. Diagnosed with stage I lung cancer or benign lesions by histologic examination;
4. Volunteered to participate in the study and signed an informed consent form.

Exclusion Criteria:

1. Previous thoracic surgery
2. Any type of chronic pain, requiring daily use of analgetics
3. Any type of chronic cough that requires daily medication
4. pregnant
5. Breast feeding
6. contraindications to NSAID
7. Combination of other tumors requiring chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient underwent a single-port thoracoscopic lung resection and had postoperative pathologic confirmation of stage I lung cancer or a benign lesion.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 12 months after surgery
  Change from baseline in pain scores on the Brief Pain Inventory and the McGill Pain Questionnaire at postoperative weeks 1, 2, 4, 12, 26, and 52.
Postoperative chronic cough | 12 months after surgery
  Number of participants with postoperative chronic cough as assessed by the Leicester Cough Questionnaire at postoperative weeks 1, 2, 4, 12, 26, and 52.
Quality of life after surgery | 12 months after surgery
  Change from baseline in quality of life scores on the European Organisation for Research and Treatment of Cancer 30 item Quality of Life Questionnaire at postoperative weeks 1, 2, 4, 12, 26, and 52.

SECONDARY OUTCOMES:
Anxiety status | 12 months after surgery
  Number of participants with anxiety as assessed by the Hospital Anxiety and Depression Scale (HADS) and the Generalized Anxiety Disorder Screener (GAD-7) at postoperative weeks 1, 2, 4, 12, 26, and 52.
Depression status | 12 months after surgery
  Number of participants with depression as assessed by the Hospital Anxiety and Depression Scale (HADS) and the Beck Depression Inventory (BDI) at postoperative weeks 1, 2, 4, 12, 26, and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Maohui Chen, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Maohui Chen, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Huang Y, Chen M, Wu Z, Liu P, Zhang S, Chen C, Zheng B. Postoperative chronic operation-related symptoms after minimally invasive lung surgery: a prospective observational protocol. BMJ Open. 2024 Aug 3;14(8):e082412. doi: 10.1136/bmjopen-2023-082412. PMID 39097304